CLINICAL TRIAL: NCT03871530
Title: A Novel Approach to Optimize Programmed Intermittent Epidural Bolus (PIEB) Delivery for Labour Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Allana, Principle Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1023951
Record Dates: First submitted 2019-03-01; First posted 2019-03-12 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Labor Pain
Keywords: Analgesia; Epidural; Labor; Obstetric Analgesia; Obstetrical
MeSH Terms: conditions — Labor Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: double-blind randomized trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Coordinate A (Experimental): PIEB "Next Bolus": 45 minutes, PIEB Interval: 50 minutes, and PIEB volume: 5 mL
  Interventions: Other: Coordinate A
- Coordinate B (Experimental): PIEB "Next Bolus": 45 minutes, PIEB Interval: 40 minutes, and PIEB volume: 6.5 mL
  Interventions: Other: Coordinate B
- Coordinate C (Experimental): PIEB "Next Bolus": 45 minutes, PIEB Interval: 50 minutes, and PIEB volume: 8 mL
  Interventions: Other: Coordinate C
- Coordinate D (Experimental): PIEB "Next Bolus": 45 minutes, PIEB Interval: 60 minutes, and PIEB volume: 6.5 mL
  Interventions: Other: Coordinate D
- Coordinate E (Experimental): PIEB "Next Bolus": 30 minutes, PIEB Interval: 40 minutes, and PIEB volume: 5 mL
  Interventions: Other: Coordinate E
- Coordinate F (Experimental): PIEB "Next Bolus": 30 minutes, PIEB Interval: 40 minutes, and PIEB volume: 8 mL
  Interventions: Other: Coordinate F
- Coordinate G (Experimental): PIEB "Next Bolus": 30 minutes, PIEB Interval: 60 minutes, and PIEB volume: 8 mL
  Interventions: Other: Coordinate G
- Coordinate H (Experimental): PIEB "Next Bolus": 30 minutes, PIEB Interval: 60 minutes, and PIEB volume: 5 mL
  Interventions: Other: Coordinate H
- Coordinate I (Experimental): PIEB "Next Bolus": 15 minutes, PIEB Interval: 50 minutes, and PIEB volume: 5 mL
  Interventions: Other: Coordinate I
- Coordinate J (Experimental): PIEB "Next Bolus": 15 minutes, PIEB Interval: 40 minutes, and PIEB volume: 6.5 mL
  Interventions: Other: Coordinate J
- Coordinate K (Experimental): PIEB "Next Bolus": 15 minutes, PIEB Interval: 50 minutes, and PIEB volume: 8 mL
  Interventions: Other: Coordinate K
- Coordinate L (Experimental): PIEB "Next Bolus": 15 minutes, PIEB Interval: 60 minutes, and PIEB volume: 6.5 mL
  Interventions: Other: Coordinate L
- Coordinate M (Experimental): PIEB "Next Bolus": 30 minutes, PIEB Interval: 50 minutes, and PIEB volume: 6.5 mL
  Interventions: Other: Coordinate M
- Coordinate N (Experimental): PIEB "Next Bolus": 30 minutes, PIEB Interval: 50 minutes, and PIEB volume: 6.5 mL
  Interventions: Other: Coordinate N

INTERVENTIONS:
Other: Coordinate A — PIEB "Next Bolus": 45 minutes, PIEB Interval: 50 minutes, and PIEB volume: 5 mL
  Arms: Coordinate A
Other: Coordinate B — PIEB "Next Bolus": 45 minutes, PIEB Interval: 40 minutes, and PIEB volume: 6.5 mL
  Arms: Coordinate B
Other: Coordinate C — PIEB "Next Bolus": 45 minutes, PIEB Interval: 50 minutes, and PIEB volume: 8 mL
  Arms: Coordinate C
Other: Coordinate D — PIEB "Next Bolus": 45 minutes, PIEB Interval: 60 minutes, and PIEB volume: 6.5 mL
  Arms: Coordinate D
Other: Coordinate E — PIEB "Next Bolus": 30 minutes, PIEB Interval: 40 minutes, and PIEB volume: 5 mL
  Arms: Coordinate E
Other: Coordinate F — PIEB "Next Bolus": 30 minutes, PIEB Interval: 40 minutes, and PIEB volume: 8 mL
  Arms: Coordinate F
Other: Coordinate G — PIEB "Next Bolus": 30 minutes, PIEB Interval: 60 minutes, and PIEB volume: 8 mL
  Arms: Coordinate G
Other: Coordinate H — PIEB "Next Bolus": 30 minutes, PIEB Interval: 60 minutes, and PIEB volume: 5 mL
  Arms: Coordinate H
Other: Coordinate I — PIEB "Next Bolus": 15 minutes, PIEB Interval: 50 minutes, and PIEB volume: 5 mL
  Arms: Coordinate I
Other: Coordinate J — PIEB "Next Bolus": 15 minutes, PIEB Interval: 40 minutes, and PIEB volume: 6.5 mL
  Arms: Coordinate J
Other: Coordinate K — PIEB "Next Bolus": 15 minutes, PIEB Interval: 50 minutes, and PIEB volume: 8 mL
  Arms: Coordinate K
Other: Coordinate L — PIEB "Next Bolus": 15 minutes, PIEB Interval: 60 minutes, and PIEB volume: 6.5 mL
  Arms: Coordinate L
Other: Coordinate M — PIEB "Next Bolus": 30 minutes, PIEB Interval: 50 minutes, and PIEB volume: 6.5 mL
  Arms: Coordinate M
Other: Coordinate N — PIEB "Next Bolus": 30 minutes, PIEB Interval: 50 minutes, and PIEB volume: 6.5 mL
  Arms: Coordinate N

SUMMARY:
Programmed intermittent epidural bolus (PIEB) for labour analgesia allows an epidural pump to be programmed to deliver small amounts of the local anesthetic and opioid solution at regularly timed intervals. However, little evidence is available to guide optimal settings for PIEB. The gaps in evidence include: (1) programmed timing for the first PIEB bolus (referred to as the "NEXT bolus") (2) determination of PIEB bolus volume (3) the interval for subsequent doses (PIEB interval). Response Surface Methodology will be utilized to best estimate the optimal PIEB settings (NEXT bolus interval, PIEB interval time, PIEB volume) by using the following clinical primary outcome measures: maternal satisfaction score, need for a clinician administered rescue bolus, and the ratio of PCEA boluses requested/delivered.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous,
* English speaking
* 18-45 years
* single gestation ≥ 37 weeks
* vertex presentation
* American Society of Anesthesiologists (ASA) Physical Status II (mild and controlled systemic disease and/or pregnancy)
* requesting an epidural for labour analgesia
* cervical dilation ≤ 7 cm at the time of initiation of epidural analgesia.

Exclusion Criteria:

* Preeclampsia or HELLP syndrome
* maternal cardiac disease
* severe or uncontrolled maternal systemic disease
* contraindication to neuraxial analgesia (i.e. coagulopathy, infection, neuropathy)
* abnormal spinal anatomy (i.e. severe scoliosis, spina bifida, spinal instrumentation)
* chronic analgesic use
* a physical or psychiatric condition which may impair cooperation
* known fetal anomalies/intrauterine fetal demise
* height < 5'0"
* Body Mass Index > 45 kg/m2

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Maternal satisfaction score | 24 hours following delivery
  quantified as 0-100, where 0 - not satisfied, and 100 - completely satisfied
Number of clinician administered rescue boluses | Start of labour epidural to delivery time
  Recorded from the Innovian anesthesia database, IntelliSpace Perinatal, or CADD®-Solis Epidural Pump
Ratio of the number of PCEA boluses requested to the number of PCEA boluses delivered | Start of labour epidural to delivery time
  Recorded on the CADD®-Solis Epidural Pump during labour and downloaded by research coordinator after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munro A, George RB, Andreou P. An Innovative Approach to Determine Programmed Intermittent Epidural Bolus Pump Settings for Labor Analgesia: A Randomized Controlled Trial. Anesth Analg. 2024 Sep 1;139(3):545-554. doi: 10.1213/ANE.0000000000006813. Epub 2024 Aug 16. PMID 38905148

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03871530/Prot_SAP_001.pdf